CLINICAL TRIAL: NCT06526169
Title: Assessment of Human Exposure to Chemical Hazards and Their Association With Food Consumption in the Singapore Population
Brief Title: Assessment of Human Exposure to Chemical Hazards
Status: Active, not recruiting | Type: Observational
Sponsor: National University of Singapore (Other)
Collaborators: Singapore Food Agency (Unknown)
Responsible Party: Principal Investigator, Mei Hui Liu, Senior Lecturer, National University of Singapore
Other Study IDs: NUS-IRB-2024-128
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Dietary Exposure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Plasma and serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ethnicity: Chinese
  Interventions: Other: Food Frequency, Social, Lifestyle, Demographic Questionnaires and Blood Collection
- Ethnicity: Malay
  Interventions: Other: Food Frequency, Social, Lifestyle, Demographic Questionnaires and Blood Collection
- Ethnicity: Indian
  Interventions: Other: Food Frequency, Social, Lifestyle, Demographic Questionnaires and Blood Collection

INTERVENTIONS:
Other: Food Frequency, Social, Lifestyle, Demographic Questionnaires and Blood Collection — Questionnaires on food frequency, social, lifestyle, and demographics will be administered to participants and will be correlated with the presence of chemical hazards in the blood. The chemical hazards analyzed will be referenced from Singapore's Total Diet Study, based on the prioritized chemical hazards of interest to investigate the distribution of risk in the population.

SUMMARY:
The aim of this study is to evaluate the occurrence of chemical hazards exposure in the Singapore population and assess their association with food consumption.

DETAILED DESCRIPTION:
Human biomonitoring is an exposure assessment approach with the potential value-add supplementation to existing sources of information for regulatory risk assessments and for supporting food safety policies. The collaboration involving academic partners from the sciences and public health disciplines to quantify the in vivo chemical exposure of chemicals will take reference from the findings in the Singapore's total diet study on the prioritised chemical hazards of interest for a more precise assessment of the distribution of risk in the population. Direct measurement of chemicals and/or metabolites in biological specimens obtained from study subjects will be conducted to provide a more comprehensive understanding on the baseline dietary chemical exposure in the local population. Dietary assessment using food frequency questionnaire will be administered to the same group of study subjects to associate human exposure to chemical hazards with food consumption across the different population groups in Singapore.

ELIGIBILITY:
Inclusion Criteria:

* Must be English-literate and able to give informed consent in English
* 21 to 60 years of age (inclusive) at screening
* Healthy adults
* Race must be Chinese or Indian or Malay
* Reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures

Exclusion Criteria:

* Known or ongoing psychiatric disorders within 3 years
* Being diagnosed with cancer, heart disease, stroke, renal failure, serious mental or physical illnesses at the time of recruitment
* Have donated blood of more than 500 mL within 4 weeks of study enrolment

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults in the Singapore population
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-08-21 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Chemical hazards occurrence | 3 years
  To evaluate the occurrence of chemical hazards exposure in the Singapore population and assess their association with food consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Mei Hui Liu, Principal Investigator — National University of Singapore
Locations (2):
- Singapore (2):
  - National University of Singapore, Singapore
  - National University of Singapore, Department of Food Science & Technology, Singapore